CLINICAL TRIAL: NCT00972842
Title: Phase I/II Trial of Lenalidomide in Combination With Vorinostat and Dexamethasone as Therapy in Relapsed or Refractory Patients With Peripheral T-Cell Non-Hodgkin's Lymphoma (PTCL)
Brief Title: Lenalidomide, Vorinostat and Dexamethasone in Relapsed Patients With Peripheral T-Cell Non-Hodgkin's Lymphoma (PTCL)
Acronym: LenVoDex
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_PTCL1; EudraCT 2008-006919-20
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Peripheral T-Cell Non-Hodgkin's Lymphoma
Keywords: PTCL; Peripheral T-Cell Non-Hodgkin's Lymphoma; Vorinostat; Lenalidomid
MeSH Terms: interventions — Vorinostat; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vorinostat, Lenalidomide — Lenalidomide: Dose escalation 10 /15 /20 /25mg/d d1-21 q28d; for 6 treatment cycles
  Vorinostat: 400 mg d1-21 q28d, for 6 treatment cycles
  Other Names: Revlimid®; Zolinza®

SUMMARY:
A standard therapy is neither established in first-line patients nor in relapsed patients with PTCL, and there is still an unmet medical need to identify novel efficacious and safe therapy regimens.

The aim of this study is to evaluate the potential of a Lenalidomide plus Vorinostat and Dexamethasone combination therapy as an effective and safe therapeutic regimen, in the treatment of relapsed PTCL following failure of prior regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed PTCL according to WHO criteria who have received max. two previous treatments for PTCL
* Age ≥ 18 years.
* Adequate bone marrow function i.e. absolute neutrophile count of > 1000/µl and thrombocytes > 75,000/µl.
* Alkaline phosphatase and transaminases ≤ 2,5 x upper limit of normal (ULN)
* Total bilirubin ≤ 2,5 x ULN
* Creatinine clearance ≥ 50 ml/min
* Female subjects of childbearing potential† must: Understand that the study medication could have an expected teratogenic risk and agree to use, and be able to comply with, effective contraception and agree to have a medically supervised pregnancy test
* Male subjects must agree to use condoms and agree not to donate semen

Exclusion Criteria:

* Prior history of malignancies, other than PTCL, unless the subject has been free of the disease for ≥ 3 years
* Prior allogeneic bone marrow transplant or plans to undergo autologous/ allogeneic bone marrow transplant within 4 weeks of the initiation of vorinostat administration
* Prior treatment with a HDAC inhibitor
* Prior treatment with Lenalidomide (patients previously treated with Thalidomide may be enrolled)
* Known history of Deep Vein Thrombosis (DVT) and/ or pulmonary embolism (PE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the maximum tolerated dose (MTD) of a Lenalidomide, Vorinostat, and Dexamethasone combination regimen in terms of occurrence of dose-limiting toxicities (DLT) at any dose level. | 6 months

SECONDARY OUTCOMES:
Remission rate of a combination therapy with Lenalidomide, Vorinostat, and Dexamethasone in a treatment refractory or relapsed population, defined as the percentage of patients achieving a complete response (CR) or partial response (PR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Hopfinger, MD, Principal Investigator — Hanusch Krankenhaus Wien
Locations (5):
- Austria (5):
  - Medizinische Universitaet Innsbruck, Abtlg. f. Haematologie und Onkologie, Innsbruck, Tyrol
  - Krankenhaus der Elisabethinen Linz, Linz
  - Krankenhaus der Stadt Linz, Linz
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - Hanusch Krankenhaus, Vienna